CLINICAL TRIAL: NCT03301467
Title: A Randomized, Double Blind, Placebo Controlled Phase 2 Study to Evaluate the Safety and Efficacy of Avacopan (CCX168) in Patients With C3 Glomerulopathy
Brief Title: Controlled Trial Evaluating Avacopan in C3 Glomerulopathy
Acronym: ACCOLADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL011_168; 1R01FD006342-01 (FDA)
Record Dates: First submitted 2017-09-22; First posted 2017-10-04 (Actual); Results first posted 2022-10-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: C3 Glomerulopathy (C3G)
Keywords: C3 Glomerulonephritis; C3 glomerulopathy; C3G; DDD; dense deposit disease; membranoproliferative glomerulonephritis; MPGN; C3GN; idiopathic MPGN
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — avacopan

STUDY DESIGN:
Intervention Model Description: Placebo crossover to active
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avacopan (Experimental): Avacopan (formerly CCX168) 10 mg capsules x 3 administered twice daily during the blinded 26 week blinded treatment period
  Interventions: Drug: Avacopan
- Avacopan Matching Placebo (Placebo Comparator): Matching placebo capsules x 3 administered twice daily during the 26 week blinded treatment period period
  Interventions: Drug: Avacopan Matching Placebo

INTERVENTIONS:
Drug: Avacopan — Orally administered
  Other Names: CCX168
  Arms: Avacopan
Drug: Avacopan Matching Placebo — avacopan matching placebo
  Other Names: placebo
  Arms: Avacopan Matching Placebo

SUMMARY:
The aim of this trial is to evaluate the effect of avacopan treatment on renal disease activity in patients with complement component 3 glomerulopathy (C3G). Funding Source - FDA OOPD

DETAILED DESCRIPTION:
C3 glomerulopathy (C3G) is characterized by evidence of alternative complement activation based on C3 deposition in the glomeruli. There are two forms of the disease: dense deposit disease (DDD) and C3 glomerulonephritis (C3GN). There is no approved treatment for patients with C3G.

This is a randomized, double blind, placebo controlled Phase 2 study to evaluate the safety and efficacy of avacopan (CCX168) in patients with C3G. Patients receive avacopan 30mg or matching placebo orally twice-daily. The placebo-controlled treatment period is 26 weeks (182 days). This will be followed by 26 weeks during which time all patients will receive avacopan (results for this second period will be reported in due course in a follow-up publication). Thereafter, all patients will be followed for eight weeks (56 days) without study drug treatment. The primary objective is to evaluate the efficacy of avacopan compared to placebo based on histologic changes in kidney biopsies taken at baseline and after 26 weeks of treatment. The primary endpoint will be based on the percent change from baseline in the C3G Histologic Index for disease activity.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven C3G, either DDD or C3GN, with or without a renal transplant, and with the following observations upon renal biopsy taken within 12 weeks prior to screening or during screening:

   1. ≥2-levels of magnitude greater staining of C3 than any combination of IgG, IgM, IgA, kappa and lambda light chains, and C1q by immunohistochemistry, and
   2. evidence of proliferative glomerulonephritis (mesangial hypercellularity of greater than 3 mesangial cells per mesangial area and/or endocapillary hypercellularity defined as an increased number of cells within glomerular capillary lumina, causing luminal narrowing) based on light microscopy, and
   3. confirmation of the presence of electron dense deposits in the glomeruli on electron microscopy corresponding with the C3 immunofluorescence positivity;
2. Male or female subjects, aged at least 18 years; where approved, adolescents (12-17 year old) may be enrolled; female subjects of childbearing potential (i.e., those who have experienced menarche and who is not permanently sterile or postmenopausal, defined as at least 12 consecutive months with no menses without an alternative medical cause) may participate if adequate contraception is used during, and for at least the three months after study completion; Male subjects with partners of childbearing potential may participate in the study if they had a vasectomy at least 6 months prior to randomization or if adequate contraception is used during, and for at least the 3 months after study completion; Adequate contraception is defined as resulting in a failure rate of less than 1% per year (combined estrogen and progestogen [oral, intravaginal, or transdermal], or progestogen-only hormonal contraception (oral, injectable, or implantable), intra-uterine device, intra-uterine hormone releasing system, bilateral tubal occlusion, vasectomized partner, or true sexual abstinence, i.e., in line with the preferred and usual lifestyle of the subject);
3. Willing and able to give written Informed Consent and to comply with the requirements of the study protocol; written Assent and Informed Consent must be obtained from the legal guardian in accordance with regional laws or regulations for subjects 12 to 17 years of age; and
4. Judged to be otherwise fit for the study by the Investigator, based on medical history, physical examination, and clinical laboratory assessments. Subjects with clinical laboratory values that are outside of normal limits (other than those specified in the Exclusion Criteria) and/or with other abnormal clinical findings that are judged by the Investigator not to be of clinical significance, may be entered into the study.

Exclusion Criteria:

1. Pregnant or nursing;
2. Tubulointerstitial fibrosis appears to be more than 50% based on standard assessment using trichrome staining of the renal biopsy;
3. Use of eculizumab or another anti-C5 antibody within 26 weeks prior to dosing;
4. Secondary C3 disease, e.g., infection-associated disease, or associated with another systemic or autoimmune disease; presence of a monoclonal spike on serum or urine protein electrophoresis or immunofixation assay;
5. Currently on dialysis or likely will require dialysis within 7 days after screening;
6. History or presence of any form of cancer within the 5 years prior to screening, with the exception of excised basal cell or squamous cell carcinoma of the skin, or carcinoma in situ such as cervical or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis;
7. Positive hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) viral screening test indicative of acute or chronic infection;
8. Evidence of tuberculosis based on interferon γ release assay (IGRA), tuberculin purified protein derivative (PPD) skin test, or chest radiography done at screening or within 6 weeks prior to screening;
9. WBC count less than 3500/μL, or neutrophil count less than 1500/μL, or lymphocyte count less than 500/μL before start of dosing;
10. Evidence of hepatic disease; AST, ALT, alkaline phosphatase, or bilirubin >3 x the upper limit of normal before start of dosing;
11. Currently using a strong inducer of the CYP3A4 enzyme, such as carbamazepine, phenobarbital, phenytoin, rifampin, or St. John's wort;
12. Known hypersensitivity to avacopan or inactive ingredients of the avacopan capsules (including gelatin, polyethylene glycol, or Cremophor) or inability to swallow the capsules;
13. Participated in any clinical study of an investigational product within 30 days prior to screening or within 5 half-lives after taking the last dose; and
14. History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the subject at unacceptable risk for study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (43):
- United States (10):
  - Clinical Site, Palo Alto, California
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Iowa City, Iowa
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, New York, New York
  - Clinical Site, Rochester, New York
  - Clinical Site, Columbus, Ohio
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, East Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah
- Belgium (4):
  - Clinical Site, Antwerp
  - Clinical Site, Brussels
  - Clinical Site, Leuven
  - Clinical Site, Liège
- Canada (2):
  - Clinical Site, Vancouver, British Columbia
  - Clinical Site, Calgary
- Denmark (3):
  - Clinical Site, Aalborg
  - Clinical Site, Copenhagen
  - Clinical Site, Odense
- France (4):
  - Clinical Site, Boulogne-sur-Mer
  - Clinical Site, Grenoble
  - Clinical Site, Paris
  - Clinical Site, Valenciennes
- Germany (5):
  - Clinical Site, Dresden
  - Clinical Site, Essen
  - Clinical Site, Hanover
  - Clinical Site, Lübeck
  - Clinical Site, Munich
- Clinical Site, Dublin, Ireland
- Italy (5):
  - Clinical Site, Bergamo
  - Clinical Site, Bologna
  - Clinical Site, Milan
  - Clinical Site, Parma
  - Clinical Site, Roma
- Netherlands (4):
  - Clinical Site, Amsterdam
  - Groningen UMC, Groningen
  - Clinical Site, Leiden
  - Clinical Site, Nijmegen
- Spain (3):
  - Clinical Site, Barcelona
  - Clinical Site, Burela de Cabo
  - Clinical Site, Madrid
- United Kingdom (2):
  - Clinical Site, London
  - Clinical Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Bomback AS, Herlitz LC, Kedia PP, Petersen J, Yue H, Lafayette RA; ACCOLADE Study Group. Safety and Efficacy of Avacopan in Patients with Complement 3 Glomerulopathy: Randomized, Double-Blind Clinical Trial. J Am Soc Nephrol. 2025 Mar 1;36(3):487-499. doi: 10.1681/ASN.0000000526. Epub 2024 Oct 11. PMID 39392695

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Avacopan-matching placebo capsules x 3 administered twice daily during the 26 week blinded treatment period period
  Avacopan-matching placebo: Orally administered
- Avacopan Group: Avacopan (formerly CCX168) 10 mg capsules x 3 administered twice daily during the blinded 26 week blinded treatment period
  Avacopan: Orally administered
Period: Overall Study
Arm/Group | Placebo Group | Avacopan Group
Started | 29 | 28
Completed | 25 | 25
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Avacopan Group | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (17.53) | 32.2 (15.03) | 34.7 (16.39)
Age, Customized [Count of Participants; unit: Participants]
  12-17 years | 2 | 0 | 2
  18-50 years | 20 | 23 | 43
  51-65 years | 4 | 4 | 8
  >65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 3 | 5
  Netherlands | 5 | 1 | 6
  Belgium | 1 | 2 | 3
  United States | 10 | 11 | 21
  Ireland | 3 | 3 | 6
  Denmark | 1 | 1 | 2
  Italy | 1 | 0 | 1
  United Kingdom | 2 | 2 | 4
  Germany | 2 | 1 | 3
  Spain | 2 | 4 | 6
Geographic Region [Count of Participants; unit: Participants]
  North America | 12 | 14 | 26
  Rest of World | 17 | 14 | 31
Age at Diagnosis of C3G [Mean (Standard Deviation); unit: years] — C3G=C3 Glomerulopathy
  years | 33.3 (17.95) | 28.2 (17.08) | 30.8 (17.56)
C3GN or DDD [Count of Participants; unit: Participants] — C3GN=C3 Glomerulonephritis; DDD=Dense Deposit
  Missing refers to one subject for whom disease type (C3GN vs DDD) could not be determined and subject was randomized in error.
  Participants
    C3GN | 25 | 23 | 48
    DDD | 4 | 4 | 8
    Missing | 0 | 1 | 1
History of Kidney Transplant [Count of Participants; unit: Participants] — Missing refers to one subject for whom disease type (C3GN vs DDD) could not be determined and subject was randomized in error.
  Participants
    Yes | 2 | 1 | 3
    No | 27 | 26 | 53
    Missing | 0 | 1 | 1
C5b-9 Stratum [Count of Participants; unit: Participants] — C5b-9 levels <= 244 ng/mL were normal according to the central laboratory used for the study. Defined by assay normal range.
  Participants
    > 244 ng/mL | 22 | 21 | 43
    <= 244 ng/mL | 7 | 7 | 14
Duration of C3G [Mean (Standard Deviation); unit: months] — Calculated from the time of first diagnosis based on renal biopsy. C3G=C3 glomerulopathy
  months | 46.7 (43.78) | 48.2 (46.38) | 47.4 (44.68)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m²] — eGFR=estimated Glomerular Filtration Rate
  mL/min/1.73m² | 72.34 (43.509) | 79.29 (39.751) | 75.75 (41.480)
UPCR [Mean (Standard Deviation); unit: g/g] — UPCR=Urine Protein to Creatinine Ratio
  g/g | 2.80 (2.435) | 4.11 (3.380) | 3.44 (2.985)
UPCR (g/g) [Count of Participants; unit: Participants] — UPCR=Urine Protein to Creatinine Ratio
  Urine protein-to-creatinine ratio (UPCR): UPCR was calculated by dividing the level of protein in a spot urine test by the creatinine level. UPCR estimates the 24-hour protein excretion in grams per day and is used in clinical practice and clinical trials to measure the severity of proteinuria in patients.
  Participants
    > 1 g/g | 21 | 22 | 43
    <= 1 g/g | 8 | 6 | 14
Urinary MCP-1:Creatinine Ratio [Mean (Standard Deviation); unit: pg/mg Creatinine] — Population: 2 patients missed baseline Urinary MCP-1 data.
  pg/mg Creatinine
    number analyzed (Participants) | 28 | 27 | 55
    (all) | 750.29 (492.542) | 1215.88 (1303.359) | 978.85 (997.191)
Body Weight [Mean (Standard Deviation); unit: kilogram(s)] | 72.65 (12.631) | 78.33 (19.229) | 75.44 (16.317)
Height [Mean (Standard Deviation); unit: centimeter(s)] | 171.41 (8.773) | 173.82 (10.805) | 172.60 (9.810)
BMI [Mean (Standard Deviation); unit: kilogram(s)/square meter] — BMI=Body Mass Index
  kilogram(s)/square meter | 24.65 (3.410) | 26.05 (6.375) | 25.34 (5.090)
EQ-5D-5L Index Score [Mean (Standard Deviation); unit: units on a scale] — EQ-5D-5L=EuroQuality of Life-5 Domains-5 Levels
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers given can be converted into an Index Score ranging from 0 for death to 1 for perfect health.
  units on a scale | 0.88 (0.145) | 0.87 (0.116) | 0.88 (0.130)
EQ-5D-5L VAS Score [Mean (Standard Deviation); unit: units on a scale] — EQ-5D-5L=EuroQuality of Life-5 Domains-5 Levels
  VAS=Visual Analog Scale
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D questionnaire includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst imaginable health) to 100 (the best imaginable health).
  units on a scale | 78.83 (20.604) | 73.61 (19.070) | 76.26 (19.862)
Viral Test Results HIV-1/2 Antibody [Count of Participants; unit: Participants] — HIV=Human Immunodeficiency Virus
  Participants
    Reactive | 0 | 0 | 0
    Non-reactive | 29 | 28 | 57
Viral Test Results - Hepatitis B Virus Surface Antigen [Count of Participants; unit: Participants]
  Reactive | 0 | 0 | 0
  Non-reactive | 29 | 28 | 57
Viral Test Results - Hepatitis C Virus Antibody [Count of Participants; unit: Participants]
  Reactive | 0 | 1 | 1
  Non-reactive | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in the C3G Histologic Index for Disease Activity - Subjects With Elevated C5b-9
Description: Change from baseline to Week 26 in the biopsy-based C3G Histologic Index for disease activity - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  C3G Histological Index for Disease Activity Scores can range from 0 to 21. A decrease indicates improvement.
  C3G=C3 glomerulopathy
Time Frame: Week 26
Population: Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat (ITT) Population. The number of subjects with data at baseline and the specified visit is reported.
  ITT Population: The ITT Population included all randomized subjects who received at least one dose of study medication; subjects with a histologic activity score of 0 at baseline or who were ongoing and had not completed the Week 26 visit were not included in the ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 21 | 19
score on a scale | -0.9 [-2.2 to 0.4] | -1.0 [-2.3 to 0.4]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.9670, ANCOVA; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-1.9 to 1.8]

2. Primary Outcome: Percent Change From Baseline to Week 26 in the C3G Histologic Index for Disease Activity - Combined C5b-9 Strata
Description: Percent change from baseline to Week 26 in the biopsy-based C3G Histologic Index for disease activity - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  C3G Histological Index for Disease Activity Scores can range from 0 to 21. A decrease indicates improvement.
  C3G=C3 glomerulopathy
  * Multiple Imputation: Missing Week 26 values are imputed using the regression method to create 100 complete datasets.
Time Frame: Week 26
Population: Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat (ITT) Population
  ITT Population: The ITT Population included all randomized subjects who received at least one dose of study medication; subjects with a histologic activity score of 0 at baseline or who were ongoing and had not completed the Week 26 visit were not included in the ITT population.
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 26 | 26
Percentage change | 26.20 (47.302) | -5.77 (5.904)
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.3083, Van Elteren's Test; Mean Difference (Final Values) = 1.02 — Test for normality showed that mean change and mean percent change were not normally distributed. As per SAP, Van Elteren's test was then applied to test mean percent change. SAP=Statistical Analysis Protocol

3. Secondary Outcome: Proportion of Subjects Who Have a Histologic Response Defined as a Decrease (Improvement) in the Biopsy-based C3G Histologic Index for Activity of at Least 35% From Baseline to 26 Weeks - Subjects With Elevated C5b-9
Description: Proportion of subjects who have a histologic response defined as a decrease (improvement) in the biopsy-based C3G Histologic Index for activity of at least 35% from baseline to 26 weeks - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  C3G Histological Index for Disease Activity Scores can range from 0 to 21. A decrease indicates improvement.
  C3G=C3 glomerulopathy
Time Frame: Week 26
Population: Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat (ITT) Population. The number of subjects with C3G Histological Index of Disease Activity Percent Change at Week 26 is reported.
  ITT Population: The ITT Population included all randomized subjects who received at least one dose of study medication; subjects with a histologic activity score of 0 at baseline or who were ongoing and had not completed the Week 26 visit were not included in the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 20 | 18
Participants
  Responder | 4 | 2
  Non-Responder | 16 | 16
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.4591, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel chi square general association statistic

4. Secondary Outcome: Proportion of Subjects Who Have a Histologic Response Defined as a Decrease (Improvement) in the Biopsy-based C3G Histologic Index for Activity of at Least 35% From Baseline to 26 Weeks - Combined C5b-9 Strata
Description: Proportion of subjects who have a histologic response defined as a decrease (improvement) in the biopsy-based C3G Histologic Index for activity of at least 35% from baseline to 26 weeks - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  C3G Histological Index for Disease Activity Scores can range from 0 to 21. A decrease indicates improvement.
  C3G=C3 glomerulopathy
Time Frame: Week 26
Population: Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat (ITT) Population. The number of subjects with C3G Histological Index of Disease Activity Percent Change at Week 26 is reported.
  The ITT Population included all randomized subjects who received at least one dose of study medication; subjects with a histologic activity score of 0 at baseline or who were ongoing and had not completed the Week 26 visit were not included in the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 25 | 25
Participants
  Responder | 7 | 4
  Non-Responder | 18 | 21
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.3106, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel chi square general association statistic

5. Secondary Outcome: Change From Baseline to Week 26 in the C3G Histologic Index for Disease Chronicity - Subjects With Elevated C5b-9
Description: Change from baseline to Week 26 in the biopsy-based C3G Histologic Index for disease chronicity over the placebo-controlled treatment period - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  C3G Histological Index for Disease Chronicity Scores can range from 0 to 10. A decrease indicates improvement.
  C3G=C3 glomerulopathy
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 21 | 19
score on a scale | 1.5 [0.9 to 2.2] | 1.1 [0.3 to 1.8]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.3368, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.5 to 0.5]

6. Secondary Outcome: Change From Baseline to Week 26 in the C3G Histologic Index for Disease Chronicity - Combined C5b-9 Strata
Description: Change from baseline to Week 26 in the biopsy-based C3G Histologic Index for disease chronicity over the placebo-controlled treatment period - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  C3G Histological Index for Disease Chronicity Scores can range from 0 to 10. A decrease indicates improvement.
  C3G=C3 glomerulopathy
Time Frame: Week 26
Population: Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat (ITT) Population. The number of subjects with data at baseline and the specified visit is reported.
  ITT Population: The ITT Population included all randomized subjects who received at least one dose of study medication; subjects with a histologic activity score of 0 at baseline or who were ongoing and had not completed the Week 26 visit were not included in the ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 26 | 26
score on a scale | 1.6 [1.1 to 2.2] | 0.8 [0.2 to 1.4]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.0401, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.7 to -0.0]

7. Secondary Outcome: Renal Function as Assessed by Percent Change From Baseline Over 26 Weeks in eGFR - Subjects With Elevated C5b-9
Description: The percent change from baseline over 26 weeks in estimated Glomerular Filtration Rate (eGFR) - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 20 | 18
Percentage change | -4.73 [-12.29 to 2.83] | 6.11 [-1.86 to 14.08]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.0534, Mixed Models Analysis; Mixed model repeated measures models with treatment group, visit, and treatment-by-visit interaction as factors and baseline as a covariate; Mean Difference (Final Values) = 10.84, 95% CI 2-sided [-0.16 to 21.85]

8. Secondary Outcome: Renal Function as Assessed by Percent Change From Baseline Over 26 Weeks in eGFR - Combined C5b-9 Strata
Description: The percent change from baseline over 26 weeks in estimated Glomerular Filtration Rate (eGFR) - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
Time Frame: Week 26
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 25 | 25
Percentage change | -5.88 [-12.32 to 0.56] | 4.79 [-1.66 to 11.23]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.0221, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 10.67, 95% CI 2-sided [1.56 to 19.78]

9. Secondary Outcome: Renal Function as Assessed by Change From Baseline Over 26 Weeks in eGFR - Subjects With Elevated C5b-9
Description: The change from baseline over 26 weeks in estimated Glomerular Filtration Rate (eGFR) - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 20 | 18
mL/min/1.73m^2 | -3.57 [-8.43 to 1.29] | 0.44 [-4.69 to 5.56]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.2638, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 4.00, 95% CI 2-sided [-3.08 to 11.08]

10. Secondary Outcome: Renal Function as Assessed by Change From Baseline Over 26 Weeks in eGFR - Combined C5b-9 Strata
Description: The change from baseline over 26 weeks in estimated Glomerular Filtration Rate (eGFR) - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
Time Frame: Week 26
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 25 | 25
mL/min/1.73m^2 | -3.35 [-7.56 to 0.85] | 0.47 [-3.75 to 4.68]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.2069, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 3.82, 95% CI 2-sided [-2.14 to 9.77]

11. Secondary Outcome: Percent Change From Baseline Over 26 Weeks in UPCR in Patients With Abnormal UPCR at Baseline - Subjects With Elevated C5b-9
Description: Percent change from baseline Over 26 Weeks in UPCR in patients with Abnormal UPCR at Baseline (>= 0.15 g/g) - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  LSM=Least Squares Mean; UPCR = Urine Protein : Creatinine Ratio
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 20 | 18
Percentage change | -14 [-34 to 12] | -16 [-36 to 12]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.9284, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; LSM UPCR Ratio = 0.98, 95% CI 2-sided [0.67 to 1.45] — LSM UPCR Ratio Week 26 vs Baseline, Avacopan:Placebo

12. Secondary Outcome: Percent Change From Baseline Over 26 Weeks in UPCR in Patients With Abnormal UPCR at Baseline - Combined C5b-9 Strata
Description: Percent change from baseline Over 26 Weeks in UPCR in patients with Abnormal UPCR at Baseline (>= 0.15 g/g) - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  LSM=Least Squares Mean; UPCR = Urine Protein : Creatinine Ratio
Time Frame: Week 26
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 25 | 24
Percentage change | -14 [-33 to 10] | -26 [-42 to -6]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.3778, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; LSM UPCR Ratio = 0.86, 95% CI 2-sided [0.60 to 1.21] — LSM UPCR Ratio Week 26 vs Baseline, Avacopan:Placebo

13. Secondary Outcome: Percent Change From Baseline Over 26 Weeks in Urinary MCP-1 - Subjects With Elevated C5b-9
Description: Percent change from baseline over 26 weeks in urinary MCP-1: creatinine ratio - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  LSM=Least Squares Mean; MCP-1=Monocyte Chemoattractant Protein-1
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 19 | 17
Percentage change | 1 [-18 to 25] | -23 [-39 to -4]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.0810, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; LSM MCP-1 Ratio = 0.76, 95% CI 2-sided [0.55 to 1.04] — LSM MCP-1 Ratio Week 26 vs Baseline, Avacopan:Placebo

14. Secondary Outcome: Percent Change From Baseline Over 26 Weeks in Urinary MCP-1 - Combined C5b-9 Strata
Description: Percent change from baseline over 26 weeks in urinary MCP-1: creatinine ratio - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  LSM=Least Squares Mean; MCP-1=Monocyte Chemoattractant Protein-1
Time Frame: Week 26
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 24 | 23
Percentage change | 1 [-17 to 23] | -12 [-28 to 7]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; Test type: Superiority; p = 0.3233, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; LSM MCP-1 Ratio = 0.87, 95% CI 2-sided [0.66 to 1.15] — LSM MCP-1 Ratio Week 26 vs Baseline, Avacopan:Placebo

15. Secondary Outcome: Change From Baseline Over 26 Weeks in EQ-5D-5L Health Scale VAS and Index Score - Subjects With Elevated C5b-9
Description: Change from baseline over 26 weeks in EQ-5D-5L Health Scale VAS and Index Score - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  EQ-5D-5L: EuroQuality of Life-5 Domains-5 Levels. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers given can be converted into an Index Score ranging from 0 for death to 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 20 | 18
score on a scale
  EQ-5D-5L VAS Score | -3.5 [-7.8 to 0.8] | -1.9 [-6.4 to 2.7]
  EQ-5D-5L Index Score | 0.0220 [-0.0206 to 0.0647] | -0.0202 [-0.0653 to 0.0249]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.6025, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-4.6 to 7.9]
Statistical Analysis 2: Comparison: Placebo Group vs Avacopan Group; EQ-5D-5L Index Score; Test type: Superiority; p = 0.1797, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.0422, 95% CI 2-sided [-0.1043 to 0.0198]

16. Secondary Outcome: Change From Baseline Over 26 Weeks in EQ-5D-5L Health Scale VAS and Index Score - Combined C5b-9 Strata
Description: Change from baseline over 26 weeks in EQ-5D-5L Health Scale VAS and Index Score - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  EQ-5D-5L: EuroQuality of Life-5 Domains-5 Levels. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers given can be converted into an Index Score ranging from 0 for death to 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: Week 26
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 25 | 25
score on a scale
  EQ-5D-5L VAS Score | 0.1 [-3.9 to 4.2] | -1.9 [-6.0 to 2.2]
  EQ-5D-5L Index Score | 0.0060 [-0.0334 to 0.0454] | -0.0138 [-0.0533 to 0.0256]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.4898, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-7.9 to 3.8]
Statistical Analysis 2: Comparison: Placebo Group vs Avacopan Group; EQ-5D-5L Index Score; Test type: Superiority; p = 0.4826, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.0199, 95% CI 2-sided [-0.0757 to 0.0360]

17. Secondary Outcome: Change From Baseline Over 26 Weeks in SF-36 v2 - Subjects With Elevated C5b-9
Description: Change from baseline over 26 weeks in SF-36 v2 - Subjects with Elevated C5b-9 (> 244 ng/mL) in the Intent-to-Treat Population.
  SF-36v2: Medical Outcomes Survey Short Form-36 version 2.
  SF-36v2 measures each of the following eight health domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Scores on each item are summed and averaged. The SF-36v2 component domain scores range from 0 (worst health) to 100 (best health).
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 21 | 19
score on a scale
  SF-36v2: Physical Functioning: number analyzed (Participants) | 20 | 18
  SF-36v2: Physical Functioning | 2.8518 [-3.2409 to 8.9446] | 3.2197 [-3.3108 to 9.7502]
  SF-36v2: Role-Physical: number analyzed (Participants) | 20 | 18
  SF-36v2: Role-Physical | -4.2592 [-11.5984 to 3.0801] | 3.5162 [-4.2634 to 11.2958]
  SF-36v2: Bodily Pain: number analyzed (Participants) | 20 | 17
  SF-36v2: Bodily Pain | 3.6 [-4.2 to 11.4] | -3.5 [-12.0 to 4.9]
  SF-36v2: General Health Perceptions: number analyzed (Participants) | 19 | 18
  SF-36v2: General Health Perceptions | -0.9 [-7.0 to 5.2] | 1.6 [-4.8 to 8.0]
  SF-36v2: Vitality: number analyzed (Participants) | 20 | 18
  SF-36v2: Vitality | -2.472 [-8.906 to 3.963] | 3.898 [-2.978 to 10.774]
  SF-36v2: Social Functioning: number analyzed (Participants) | 20 | 17
  SF-36v2: Social Functioning | 4.58 [-2.30 to 11.47] | 0.34 [-7.20 to 7.88]
  SF-36v2: Role-Emotional: number analyzed (Participants) | 20 | 18
  SF-36v2: Role-Emotional | 0.6859 [-6.8507 to 8.2225] | 3.2461 [-4.6899 to 11.1821]
  SF-36v2: Mental Health: number analyzed (Participants) | 20 | 18
  SF-36v2: Mental Health | 2.423 [-3.684 to 8.530] | 2.730 [-3.791 to 9.251]
  SF-36v2: Physical Component | -0.3257 [-2.6090 to 1.9576] | 0.0762 [-2.4423 to 2.5947]
  SF-36v2: Mental Component | 0.7556 [-2.3560 to 3.8672] | 0.7608 [-2.6341 to 4.1558]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; SF-36v2: Physical Component Score; Test type: Superiority; p = 0.8161, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.4019, 95% CI 2-sided [-3.0402 to 3.8440]
Statistical Analysis 2: Comparison: Placebo Group vs Avacopan Group; SF-36v2: Mental Component Score; Test type: Superiority; p = 0.9982, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.0052, 95% CI 2-sided [-4.5994 to 4.6099]

18. Secondary Outcome: Change From Baseline Over 26 Weeks in SF-36 v2 - Combined C5b-9 Strata
Description: Change from baseline over 26 weeks in SF-36 v2 - Combined C5b-9 Strata (elevated [> 244 ng/mL] and non-elevated C5b-9) in the Intent-to-Treat Population.
  SF-36v2: Medical Outcomes Survey Short Form-36 version 2.
  SF-36v2 measures each of the following eight health domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Scores on each item are summed and averaged. The SF-36v2 component domain scores range from 0 (worst health) to 100 (best health).
Time Frame: Week 26
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 26 | 26
score on a scale
  SF-36v2: Physical Functioning: number analyzed (Participants) | 25 | 25
  SF-36v2: Physical Functioning | 2.9619 [-2.7150 to 8.6389] | 4.6532 [-1.1123 to 10.4187]
  SF-36v2: Role-Physical: number analyzed (Participants) | 25 | 25
  SF-36v2: Role-Physical | -2.4712 [-9.6179 to 4.6755] | 1.2077 [-5.9734 to 8.3887]
  SF-36v2: Bodily Pain: number analyzed (Participants) | 25 | 24
  SF-36v2: Bodily Pain | 1.5 [-5.7 to 8.7] | -2.0 [-9.3 to 5.4]
  SF-36v2: General Health Perceptions: number analyzed (Participants) | 24 | 25
  SF-36v2: General Health Perceptions | -1.0 [-6.6 to 4.6] | 0.7 [-4.9 to 6.2]
  SF-36v2: Vitality: number analyzed (Participants) | 25 | 25
  SF-36v2: Vitality | -0.468 [-6.283 to 5.348] | 4.085 [-1.782 to 9.952]
  SF-36v2: Social Functioning: number analyzed (Participants) | 25 | 24
  SF-36v2: Social Functioning | 4.66 [-1.41 to 10.73] | 1.55 [-4.66 to 7.76]
  SF-36v2: Role-Emotional: number analyzed (Participants) | 25 | 25
  SF-36v2: Role-Emotional | 4.3024 [-3.3147 to 11.9195] | 7.8375 [0.2129 to 15.4620]
  SF-36v2: Mental Health: number analyzed (Participants) | 25 | 25
  SF-36v2: Mental Health | 1.503 [-3.911 to 6.917] | 3.914 [-1.543 to 9.370]
  SF-36v2: Physical Component | -0.3578 [-2.5452 to 1.8296] | -0.5096 [-2.7680 to 1.7489]
  SF-36v2: Mental Component | 1.3591 [-1.7970 to 4.5153] | 2.3874 [-0.8529 to 5.6277]
Statistical Analysis 1: Comparison: Placebo Group vs Avacopan Group; SF-36v2: Physical Component Score; Test type: Superiority; p = 0.9242, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.1518, 95% CI 2-sided [-3.3192 to 3.0156]
Statistical Analysis 2: Comparison: Placebo Group vs Avacopan Group; SF-36v2: Mental Component Score; Test type: Superiority; p = 0.6534, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.0283, 95% CI 2-sided [-3.4972 to 5.5537]

19. Secondary Outcome: Number of Subjects With Treatment-emergent SAEs, AEs, Relatedness to Study Medication and Withdrawals Due to AEs
Description: Number of Subjects with Treatment-emergent SAEs, AEs, relatedness to study medication and Withdrawals Due to AEs
  AEs=Adverse events SAEs=Serious adverse events TEAE=Treatment-emergent adverse events 'Possibly related' refers to the Investigators' causality assessment
Time Frame: From day 1 throughout the study period (day 182/week 26)
Population: Safety Population: The safety population included all subjects who were randomized and had received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 29 | 28
participants
  Number of subjects with at least one TEAE | 24 | 25
  Number of subjects with SAEs | 3 | 3
  Number of subjects with TEAEs possibly related to Study Medication | 11 | 10
  Number of subjects with TEAEs leading to discontinuation | 1 | 1

20. Secondary Outcome: Number of Treatment-emergent SAEs, AEs, Relatedness to Study Medication and Withdrawals Due to AEs
Description: Number of Treatment-emergent SAEs, AEs, relatedness to study medication and Withdrawals Due to AEs
  AEs=Adverse events SAEs=Serious adverse events TEAE=Treatment-emergent adverse events 'Possibly related' refers to the Investigators' causality assessment
Time Frame: From day 1 throughout the study period (day 182/week 26)
Population: as for outcome 19
Measure: Number; unit: Adverse events
Arm/Group | Placebo Group | Avacopan Group
Number analyzed (Participants) | 29 | 28
Adverse events
  Number of TEAEs | 107 | 149
  Number of SAEs | 4 | 6
  Number of TEAEs possibly related to Study Medication | 24 | 38
  Number of TEAEs leading to discontinuation | 2 | 2

ADVERSE EVENTS:
Time Frame: From day 1 throughout the study period (day 182/week 26)
Description: An adverse event is considered treatment-emergent if the start date/time of the event is on or after the date/time of first study drug treatment up to the final observation in the double-blind treatment period (week 26).
Groups:
- Placebo Group: Avacopan-matching placebo capsules x 3 administered twice daily during the 26 week blinded treatment period period
  Avacopan-matching placebo: Orally administered
  The safety population included all subjects who were randomized and had received at least one dose of study drug.
- Avacopan Group: Avacopan (formerly CCX168) 10 mg capsules x 3 administered twice daily during the blinded 26 week blinded treatment period
  Avacopan: Orally administered
  The safety population included all subjects who were randomized and had received at least one dose of study drug.
Arm/Group | Placebo Group | Avacopan Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/29 | 3/28
Other Adverse Events (participants affected / at risk) | 24/29 | 25/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=29) | Avacopan Group (N=28)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial parotitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=29) | Avacopan Group (N=28)
Oedema peripheral (General disorders) | 1 (1) | 5 (6)
Fatigue (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 2 (4) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3)
Nasopharyngitis (Infections and infestations) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (4)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 0 (0) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 5 (5)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 3 (4)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide Sponsor with an advance copy of any proposed publication or oral presentation at least 60 days prior to the planned date of submission or presentation and Sponsor shall have 60 days to review the proposed publication. Sponsor may request in writing, and the PI shall agree to, (a) the deletion of any Confidential Information, (b) any reasonable changes requested by Sponsor, or (c) a delay of such proposed submission for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03301467/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03301467/SAP_001.pdf